CLINICAL TRIAL: NCT06527664
Title: Innovative Technologies for Cost-Effective Healthcare Delivery for Salvage Procedures of Failed Treatments of Osteoarthritis: Specific Biomimetics Solutions to Reduce a Growing Problem With a High Social and Economic Impact.(CustomPN)
Brief Title: Innovative Technologies for Salvage Procedures of Failed Treatments of Osteoarthritis: Biomimetics Solutions (CustomPN)
Acronym: CustomPN
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: 344/2024/Oss/IOR
Record Dates: First submitted 2024-07-23; First posted 2024-07-30 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Bone Loss; Hip Prosthesis Infection; Arthroplasty Complications
Keywords: revision hip arthroplasty; custom-made implant; additive manufacturing
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Custom-made: Revision hip arthroplasty performed for non-oncological reasons, with Paprosky III bone loss
  Interventions: Device: custom-made acetabular implant

INTERVENTIONS:
Device: custom-made acetabular implant — custom-made acetabular implant produced with additive manufacturing, to fill the bony loss in Paprosky III bone defects

SUMMARY:
In this prospective multicenter study, a population of adult individuals consecutively treated for revision hips, requiring a custom-made acetabular implant for non-oncological reasons, will be included. The custom-made implant is a personalized implant produced using additive manufacturing, based on the pre-operative CT scan that details the bone damage. Patients eligible for this implant are those with severe acetabular bone damage Paprosky 3 (loss of the superolateral part and one of the two ventro-caudal walls).

Preoperatively, the patient will undergo a clinical evaluation. Data will be collected on the patient's general health status with the Charlson score, the reason for revision, number of revisions, type of implant in place, and the time elapsed between the failed implant and the revision in question. The bone deficit will be studied through CT measurements according to qualitative and quantitative scales. During the surgery, information on intraoperative complications will be collected. In the postoperative period, perioperative complications will be collected according to the Clavien Dindo classification. The clinical radiographic evaluations will be carried out during outpatient follow-up visits at 1, 3, 12, 24, and 36 months after revision. They include the Harris Hip Score clinical score, the EQ-5D PROM, and the patient's satisfaction level (qualitative assessment in 4 grades: unsatisfied, slightly satisfied, moderately satisfied, fully satisfied). The positional parameters of the implant will be evaluated, as compared to the immediate post-operative X-ray: acetabular abduction, acetabular anteversion, center of rotation height, center of rotation medialization, and inclination of the custom-made component. From 12 months onwards, the osteointegration characteristics of the component will be assessed: presence of radial trabeculae at the interface, superolateral and inferior reinforcements, stress shielding, absence of radiolucent lines. Re-revision rates will be determined using the Kaplan-Meier method. The reasons for re-revision will be noted.

DETAILED DESCRIPTION:
Osteoarthritis (OA) increased from 247.51 million people in 1990 to 527,81 million in 2019. OA places a huge burden on healthcare services accounting for 1-2,5% of the gross national products and the cost is expected to quadruple by 2030. Total joint replacement (TJR) represents the standard of care of end-stage OA. TJR is projected to nearly double by 2026. Unfortunately, TJR are subject to failure, thus the number of revision procedures is also growing, accounting for 5-6% of all TJR. Failure of TJR represents a dramatic event for patients and National Health Systems. Patients suffer enormous disability, with impact on function, emotional sphere, and loss of autonomy. The average cost of treatment is almost doubled compared to TJR, and in case of periprosthetic joint infections almost tripled. In patients under 65 years (with a failure rate of 9%-12%), the full return to work is reported only in 7%-33% of the cases, and not earlier then 1 year after the surgery, while around 50% retired or remained on welfare benefits. Current technology is not enough to overcome this set of problems, while actual projections predict a 43%-70% increase in revisions by 2030. In particular, revision hips involve various diagnoses and settings: in some cases, the severe bone loss makes the reconstruction very complex. In these cases, acetabular reconstruction can be performed with off-the-shelf implants, but outcomes are not always consistent and reproducible. Thus, in cases of severe acetabular bone loss, it may be very useful to proceed with a customized implant, designed according to the patient's needs. Implants produced in this way are designed based on the patient's pre-operative CT scan using additive manufacturing technology. The purpose is to offer a personalized bone filling of the defect with a highly porous interface that promotes osteointegration. Currently, most of the custom-made implants are performed for oncological cases. On the contrary, there are few indications on the clinical and radiological outcomes of custom-made acetabular reconstructions in revision hips with severe bone loss in non-oncological cases. The purpose of this project is to validate an innovative and reliable technology (custom-made acetabular component produced using additive manufacturing) for managing non-oncological revisions, assessing short term outcomes.

The aims are:

Description of demographic characteristics and bone defect in candidates for acetabular reconstruction with custom-made implants Perioperative complications and implant survival Clinical evaluation of custom-made implants in custom-made acetabular reconstructions in hip prosthesis revisions with severe bone loss (clinical score Harris Hip Score; subjective score PROM EQ-5D; post-operative patient satisfaction level) Radiographic evaluation (positioning and osteointegration) of custom-made implants in custom-made acetabular reconstructions in hip prosthesis revisions with severe bone loss This is a prospective multicenter study. The study population will consist of adult individuals consecutively treated for revision hips, requiring a custom-made acetabular implant. Patients with a diagnosis leading to an oncological revision will not be included. The custom-made implant is a personalized implant created by an external company based on the pre-operative CT scan that details the bone damage. Patients eligible for this implant are those with severe acetabular bone damage Paprosky 3 (loss of the superolateral part and one of the two ventro-caudal walls). In these cases, off-the-shelf therapeutic options are limited and achieve uncertain outcomes: therefore, a custom-made component with ultra-porous anchoring surfaces can represent a highly advantageous therapeutic choice. After identifying the suitable patient and obtaining their consent for the study, a pre-operative CT scan will be performed as per normal clinical practice for every revision. After uploading it to the dedicated website or app of the company, this CT scan will be used for the manufacturing of the custom-made implant by a third-party company. The company will also provide plastic phantoms for preliminary study of the implant. Upon approval of the implant production, the company will manufacture the implant according to current regulations and production techniques, following previous and established clinical practice. The device will be accompanied by personalized instrumentation, such as cutting guides, positioners, calipers, and plastic simulation phantoms, to facilitate the surgical procedure. The implant and the produced instrumentation will be delivered to the reference center after performing the patient's surgical planning.

Preoperatively, the patient will undergo an evaluation with the Harris Hip score clinical score. Additionally, data will be collected on the patient's general health status with the Charlson score, the reason for revision, number of revisions, type of implant in place, and the time elapsed between the failed implant and the revision in question. The bone deficit will be studied through CT measurements according to qualitative and quantitative scales.

During the surgery, information on intraoperative complications will be collected. In the postoperative period, perioperative complications will be collected according to the Clavien Dindo classification. The clinical radiographic evaluations will be carried out during outpatient follow-up visits at 1, 3, 12, 24, and 36 months after revision. They include the Harris Hip Score clinical score, the EQ-5D PROM, and the patient's satisfaction level (qualitative assessment in 4 grades: unsatisfied, slightly satisfied, moderately satisfied, fully satisfied). The positional parameters of the implant will be evaluated, as compared to the immediate post-operative X-ray: acetabular abduction, acetabular anteversion, center of rotation height, center of rotation medialization, and inclination of the custom-made component. From 12 months onwards, the osteointegration characteristics of the component will be assessed: presence of radial trabeculae at the interface, superolateral and inferior reinforcements, stress shielding, absence of radiolucent lines. Re-revision rates will be determined using the Kaplan-Meier method. The reasons for re-revision will be noted.

ELIGIBILITY:
Inclusion Criteria:

* need of custom-made acetabular implant on the basis of CT and X-ray evaluation ()
* pre-operative CT scan
* adults patients (minimum age: 18 years)
* complete medical charts
* patients' availability

Exclusion Criteria:

* oncological reasons for revision
* other types of revision implant (non custom)
* inadequate medical chart
* lack of pre-operative CT scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult individuals (minimum age: 18 years) consecutively treated for revision hips (non-oncological reasons) requiring a custom-made acetabular implant. Patients will be enrolled in 4 tertiary centers (multicenter prospective study). Patients eligible for this implant are those with severe acetabular bone damage Paprosky 3 (loss of the superolateral part and one of the two ventro-caudal walls).
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Perioperative complications | 0-30 days
  Clavien-Dindo classification: 5 stages with IIIA and IIIB, IV A and IV B. I stage: minimal complications, V stage: death of the patient.
Objective clinical outcomes | 0-18 months
  Harris Hip Score. Numerical scale assessing mobility, pain and functionality. Range: 0-100. 100 is the best objective outcome.
Subjective clinical outcomes | 0-18 months
  EQ-5D-5L. Subjective score with 5 dimensions: mobility, self-care, pain, usual activity, anxiety/depression (5 levels per each assessment). Weighted index on a 0-1 scale. Best outcome: 1
Subjective clinical outcomes (satisfaction) | 0-18 months
  Percentage of satisfied patients per single level. 4 levels, from not satisfied to completely satisfied.
Survival rates | 0-18 months
  Survival rates using Kaplan Meier curve. Range: 0-100%. Best outcome: 100%

SECONDARY OUTCOMES:
Osseointegration of the acetabular component | 12-18 months
  Percentages of cases with good osseointegration of the acetabular component according to Moore's criteria. At least three criteria among: presence of radial trabeculae at the interface, presence of superolateral buttress, presence of inferior buttress, presence of medial stress shielding, absence of radiolucent lines. Range: 0-100%. Best outcome: 100%

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Traina, Prof, Principal Investigator — IRCCS Istituto Ortopedico Rizzoli
Locations (1):
- Chirurgia Protesica e dei Reimpianti di Anca e Ginocchio, IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Romagnoli M, Zaffagnini M, Carillo E, Raggi F, Casali M, Leardini A, Marcheggiani Muccioli GM, Grassi A, Zaffagnini S. Custom-made implants for massive acetabular bone loss: accuracy with CT assessment. J Orthop Surg Res. 2023 Sep 30;18(1):742. doi: 10.1186/s13018-023-04230-5. PMID 37777776
- [Result] Pandey AK, Zuke WA, Surace P, Kamath AF. Management of acetabular bone loss in revision total hip replacement: a narrative literature review. Ann Jt. 2023 Oct 5;9:21. doi: 10.21037/aoj-23-23. eCollection 2024. PMID 38694811
- [Result] Jones SA, Parker J, Horner M. Can a reconstruction algorithm in major acetabular bone loss be successful in revision hip arthroplasty? Bone Joint J. 2024 May 1;106-B(5 Supple B):47-53. doi: 10.1302/0301-620X.106B5.BJJ-2023-0809.R1. PMID 38688489
- [Result] Kim K, Sandiford NA. The Role of Three-Dimensional Custom Printing in Revision Total Hip Arthroplasty. Surg Technol Int. 2023 Sep 15;42:369-373. doi: 10.52198/23.STI.42.OS1698. PMID 37675989
- [Result] Pardo F, Bordini B, Castagnini F, Giardina F, Faldini C, Traina F. Are powder-technology-built stems safe? A midterm follow-up registry study. J Mater Sci Mater Med. 2021 Jan 20;32(1):10. doi: 10.1007/s10856-020-06481-8. PMID 33471238
- [Result] Castagnini F, Mariotti F, Tassinari E, Bordini B, Zuccheri F, Traina F. lsolated acetabular revisions of articular surface replacement (ASR) XL implants with highly porous titanium cups and Delta bearings. Hip Int. 2021 Mar;31(2):250-257. doi: 10.1177/1120700019874442. Epub 2019 Sep 4. PMID 31480877

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-23): https://cdn.clinicaltrials.gov/large-docs/64/NCT06527664/Prot_SAP_000.pdf